CLINICAL TRIAL: NCT01512654
Title: Assessment of an Enhanced Version of a Personalized Glucose Predictive and Therapy Advisory System (DIAdvisor-2) for Diabetic Patients Treated by Basal-Bolus Insulin Regimens
Brief Title: Personalized Glucose Predictive and Therapy Advisory System - DIAdvisor 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 8266 3; ID-RCB : 2011-A00513-38 (Other: Afssaps)
Record Dates: First submitted 2011-09-29; First posted 2012-01-19 (Estimated); Last update posted 2021-10-20 (Actual); Status verified 2014-12

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1
Keywords: diabetes; diadvisor; type 1 diabetes; type 2 diabetes; glucose prediction; cgm prediction; algorithm; therapy advices
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- algorithm DIAdvisor activated (Other): Glucose predictions and therapy advices will be displayed to the patient. Patients will be asked to follow the advices suggested by DIAdvisor system according to their own judgement. Patient will decide his need of insulin according to the results given by the HemoCue glucometer, CGM trends, glucose predictions as well as therapy advices. In case of any doubt with the predictions displayed or the advices suggested, the patients will be invited to ask study personal and/or the study physician for help.
  Interventions: Device: Personalized Glucose Predictive and Therapy Advisory System (DIAdvisor)
- algorithm of DIAdvisor disactivated (Other): Glucosepredictions and therapy advices will not be displayed. Patient will decide his need of insulin according to the results given by the HemoCue glucometer and CGM trends. He/She will inject insulin at mealtimes or program a bolus on his/her pump by him/herself and will adapt his/her basal insulin doses or pump delivery rates as usual. As needed or on request and more particularly if hypo or hyperglycaemia occurs, the subject will be advised and helped by nurses and physicians.
  Interventions: Device: Personalized Glucose Predictive and Therapy Advisory System (DIAdvisor)

INTERVENTIONS:
Device: Personalized Glucose Predictive and Therapy Advisory System (DIAdvisor) — Glucose predictions and therapy advices will not be displayed. Patient will decide his need of insulin according to the results given by the HemoCue glucometer and CGM trends. He/She will inject insulin at mealtimes or program a bolus on his/her pump by him/herself and will adapt his/her basal insulin doses or pump delivery rates as usual. As needed or on request and more particularly if hypo or hyperglycaemia occurs, the subject will be advised and helped by nurses and physicians.
  Arms: algorithm of DIAdvisor disactivated
Device: Personalized Glucose Predictive and Therapy Advisory System (DIAdvisor) — Glucose predictions and therapy advices will be displayed to the patient. Patients will be asked to follow the advices suggested by DIAdvisor system according to their own judgement. Patient will decide his need of insulin according to the results given by the HemoCue glucometer, CGM trends, glucose predictions as well as therapy advices. In case of any doubt with the predictions displayed or the advices suggested, the patients will be invited to ask study personal and/or the study physician for help.
  Arms: algorithm DIAdvisor activated

SUMMARY:
The primary purpose of this study is to see whether a tool that predict blood glucose and suggest therapy advices can help type 1 diabetic patients.

DETAILED DESCRIPTION:
During this study, we would like to assess the efficacy in keeping blood glucose in a safe range (70-180 mg/dL) of the second generation of a Glucose Predictive and Therapy Advisory system in diabetic patients treated by basal-bolus insulin regimens using pumps or multiple daily injections. We want to compare the time spent in safe range while using the predictor and advisor outputs and when the patient is not using them. This is a randomized controlled crossover trial. Patient will come for two admissions of 3 days, one with the DIAdvisor system fully activated, and one with the prediction and advice features disabled.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be aged between 18 (inclusive) and 70 years old
2. Patients diagnosed with type 1 or type 2 diabetes according to WHO criteria for at least one year prior to study entry
3. Patient treated by a basal-bolus insulin therapy using an external pump or multiple-daily injections. The insulin regimen has to be stable for the previous six months. NPH insulin use will not be acceptable.
4. Patient should have stable diabetes with a HbA1c between ≥ 7.5 % and < 10.5 % with no keto-acidosis for the previous 6 months.
5. Patient must have a Body Mass Index (BMI) lower than 35 Kg/m²
6. Patient must be willing to undergo all study procedures
7. Patient must be affiliated or beneficiary of a social medical insurance
8. Patient has signed informed consent form prior to study entry

Exclusion Criteria:

1. Patient is pregnant, or breast feeding during the period of the study
2. Patient has impaired renal function with a creatinine blood concentration over 150 μmol/L
3. Patient has a liver disease (ALAT, ASAT > 2 x upper limit of normal range)
4. Patient is treated by sulfamides, GLP-1 analogues, DPP-IV inhibitors or glitazones
5. Alcohol or drug addiction, as identified by investigator during screening visit
6. Allergy to sensors or one of their components
7. Manifest psychological disorders
8. Patient health status is not compatible with physical exercise
9. Patient is actively enrolled in another clinical trial or was part of study within 30 days
10. Persons deprived of freedom, adults protected by law or vulnerable persons

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-09; Primary Completion 2009-02 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Percentage of total time spent by patients in safe range (70-180mg/dL) | during 3 days with DIAdvisor 2
  The primary endpoint is the percentage of total time spent by patients in safe range (70-180mg/dL). A clinically significant benefit will be reached if an increase of at least 10% of total time in range is obtained while using DIAdvisor-2.

SECONDARY OUTCOMES:
Percentage of total time spent in hypoglycemia (< 70 mg/dL) | during 3 days with DIAdvisor 2
Percentage of total of time spent in hyperglycemia (>180 mg/dL) | during 3 days with DIAdvisor 2
Mean of YSI blood glucose during total period, night time and meal periods | during the two 3 days-hospitalizations
Percentage paired glucose values | during 3 days with DIAdvisor 2
  Percentage paired glucose values: Predicted glucose t+20min vs. real glucose t to t+20min in A&B zones of EGA > 80% AND < 5% in E zone of EGA
Coherence between system advices and physician recommendations > 0.80 | during 3 days with DIAdvisor 2
Score of patient survey regarding the acceptability of DIAdvisor-2 system | during 3 days with DIAdvisor 2

CONTACTS AND LOCATIONS:
Locations (3):
- Institute for Clinical and Experimental Medicine, Prague, Czechia
- Montpellier University Hospital, Montpellier, France
- Universita Degli Studi di Padova, Padua, Italy